CLINICAL TRIAL: NCT03163654
Title: Novel Porcine Dermal Matrix Vs. Connective Tissue Graft in the Treatment of Multiple Adjacent Gingival Recessions of Miller Class I and II: a 12-month Randomized Controlled Clinical Trial
Brief Title: Novel Porcine Dermal Matrix in the Treatment of Multiple Adjacent Gingival Recessions
Acronym: NPDMMAGR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Botiss Medical AG (Other)
Responsible Party: Principal Investigator, Dragana Rakasevic, Doctor of dental medicine, University of Belgrade
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 36/24
Record Dates: First submitted 2017-05-21; First posted 2017-05-23 (Actual); Last update posted 2017-05-30 (Actual); Status verified 2017-05

CONDITIONS: Recession, Gingival
Keywords: multiple gingival recessions; collagen matrix; connective tissue graft; tunnel technique
MeSH Terms: conditions — Gingival Recession

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Participant, Investigator
Masking Description: Single Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Active Comparator): Surgery 1: The tunnel technique for covering multiple gingival recessions. Graft: porcine-derived acellular dermal collagen matrix (PADM, mucoderm® ).
  Interventions: Procedure: Surgery 1
- Control group (Active Comparator): Surgery 2: The tunnel technique for covering multiple gingival recessions. Graft: connective tissue graft
  Interventions: Procedure: Surgery 2

INTERVENTIONS:
Procedure: Surgery 1 — Following local anaesthesia (Articaine hydrochloride 4% with 1:200,000 epinephrine injection) administration, sulcular incisions were made in the recession's areas of teeth without damaging interdental papilla. Mucoperiosteal (MP) dissections were made using the periostal elevator creating the deep pouch beyond the mucogingival junction so that the (MP) flap could be moved coronally without tension. Porcine-derived acellular dermal collagen matrix (PADM) was positioned at the level of a cemento-enamel junction (CEJ) and skin tight for teeth to avoid forming a blood clot. Separate single sutures per tooth with 5-0 resorbable suture were used to stabilise graft. The tunnel flap was positioned coronally above the CEJ to completely cover the graft and sutured with non-resorbable polypropylene suture.
  Arms: Experimental group
Procedure: Surgery 2 — Following local anaesthesia (Articaine hydrochloride 4% with 1:200,000 epinephrine injection) administration, sulcular incisions were made in the recession's areas of teeth without damaging interdental papilla. Mucoperiosteal (MP) dissections were made using the periostal elevator creating the deep pouch beyond the mucogingival junction so that the (MP) flap could be moved coronally without tension. Connective tissue graft was positioned at the level of a cemento-enamel junction (CEJ) and skin tight for teeth to avoid forming a blood clot. Separate single sutures per tooth with 5-0 resorbable suture were used to stabilise graft. The tunnel flap was positioned coronally above the CEJ to completely cover the graft and sutured with non-resorbable polypropylene suture.
  Arms: Control group

SUMMARY:
The aim of this study was to assess the clinical efficacy of the acellular porcine derived collagen matrix (PADM) in comparison with connective tissue graft (SCTG ) in the treatment of multiple adjacent gingival recessions (MAGR). The primary objectives of the study were to evaluate mean and complete roots coverage. Additionally, the secondary objective was to evaluate and compare the clinical effectiveness of PADM and SCTG for the treatment of MAGR defects applying modified coronally advanced tunnel technique (MCAT).

DETAILED DESCRIPTION:
Treatment of multiple adjacent gingival recessions (MAGR) still presents a challenge for the clinician. The management of soft tissues becomes more complicated and the wound healing may be compromised by a variety of factors.

According to the available medical databases, predictable root coverage is possible for multiple-tooth recession defects using subepithelial connective tissue graft (SCTG) procedures. However, alternative materials to SCTG are supported by evidence of varying strength, with the need for additional research to confirm their performance and success rate. Because of that, the aim of this study was to assess the clinical efficacy of the acellular porcine derived collagen matrix (PADM) in comparison with connective tissue graft (SCTG ) in the treatment of multiple adjacent gingival recessions (MAGR).

This study is a randomised controlled clinical trial of 12 months duration. Sixteen patients with a total of 81 MAGR Miller's Class I or II were enrolled in this study. Recessions were randomly treated with PADM and SCTG, combined with a modified coronally advanced tunnel technique (MCAT). Several parameters, such as gingival recession coverage (RC), keratinized tissue width (KTW), keratinized tissue thickness (KTT) and clinical attachment level (CAL) were recorded at baseline and one year postoperatively. Healing index (HI) was registered on 1st, 2nd, and 3rd-week post-surgery in order to estimate healing events.

ELIGIBILITY:
Inclusion Criteria:

1. At least two multiple maxillaries or mandibular Miller's Class I and II recession, more than >2mm defects together with similar contralateral lesions
2. No active periodontal disease with PD>4mm
3. Absence of the radiographic signs of periapical infection on the teeth to be treated or on the adjacent teeth
4. A full mouth plaque index <20% and gingival index < 1

Exclusion Criteria:

1. The inflammatory periodontal disease/ Untreated periodontal conditions
2. Previous surgical attempt to correct gingival recession
3. Pregnant or breastfeeding women
4. Systemic diseases with compromised healing potential or infectious diseases

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2014-12; Primary Completion 2016-04 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
mean root coverage (MRC) | 12 months
  The percentage of covered recession area (MRC)
complete root coverage (CRC) | 12 months
  The percentage rate of patients with complete coverage of all recessions (CRC)

SECONDARY OUTCOMES:
gingival recession (GR) | 12 months
  Distance measured at the mid-buccal aspect of the tooth from the cemento-enamel junction to the most apical point of the gingival margin
gingival recession width (GRW) | 12 months
  measured at mesio-distal direction at the level of cemento-enamel junction
Keratinized tissue wide (KTW) | 12 months
  Distance from the mucogingival junction to the gingival margin
Gingival thickness (GT) | 12 months
  Measured at the mid- buccal aspect of treated tooth on the long axis
Clinical attachment level (CAL), | 12 months
  Distance from the cemento enamel junction to the deepest point of the gingival sulcus

OTHER OUTCOMES:
Probing depth (PD) | 12 months
  Distance from the gingival margin to the bottom of the sulcus

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Periodontal and Oral Mucosa Diseases, Belgrade, Serbia

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Aroca S, Keglevich T, Barbieri B, Gera I, Etienne D. Clinical evaluation of a modified coronally advanced flap alone or in combination with a platelet-rich fibrin membrane for the treatment of adjacent multiple gingival recessions: a 6-month study. J Periodontol. 2009 Feb;80(2):244-52. doi: 10.1902/jop.2009.080253. PMID 19186964